CLINICAL TRIAL: NCT02719977
Title: A Phase I Study of CX5461
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Senhwa Biosciences, Inc. (Industry); Stand Up To Cancer (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I231
Record Dates: First submitted 2016-03-21; First posted 2016-03-25 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2023-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — CX 5461

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CX-5461 (Experimental): CX5461 as intravenous infusion on day 1 and day 8 every 4 weeks. A day 1 every 3 weeks schedule may be used if the day 1 and day 8 every 4 weeks schedule is not tolerable
  Interventions: Drug: CX5461

INTERVENTIONS:
Drug: CX5461

SUMMARY:
CX5461 is a new type of drug for many types of cancer, particularly cancers that cannot easily repair damage to their cells. This may help to slow down the growth of cancer or may cause cancer cells to die. CX5461 has been shown to shrink tumours in animals and has been studied in a few people and seems promising but it is not clear if it can offer better results than standard treatment.

DETAILED DESCRIPTION:
The purpose of this study is to find the dose of a new therapy, CX5461, that can be tolerated without causing very severe side effects and to see what effects the study drug has this cancer. Participants are given CX5461 and are watched very closely to see what side effects they have and to make sure the side effects are not severe. If serious side effects are seen in patients at the first dose level, doses of CX5461 may be lowered in subsequent patients. If the side effects are not serious, then more participants are asked to join this study and are given higher doses. This will continue until a dose is found that causes severe but temporary side effects. Doses higher than that will not be given.

ELIGIBILITY:
Inclusion Criteria:

- Tumour Type Phase I Escalation: Patients must have histologically/and or cytologically confirmed solid malignancy that is advanced/metastatic/recurrent or unresectable and for which no curative therapy exists.

Phase I Expansion: Patients must have metastatic/recurrent/locally advanced/unresectable breast cancer with known BRCA1/2 or HRD germline aberrations.

* All patients must have a formalin fixed paraffin embedded tissue block (from primary or metastatic tumour) available and must have provided informed consent for the release of the block. All patients must also have provided informed consent for a whole blood sample (after implementation of amendment 3).
* All patients enrolled after the implementation of Amendment 2 must also have provided informed consent for, and be willing to undergo, a skin biopsy (of an area including hair follicles, that is not sun-exposed) prior to treatment (after registration) and after cycle 1 day 15 (C1D16). Paired tumour biopsies will also be required for 6-8 patients enrolled to the RP2D expansion. Note: During accrual to this portion of the study, it may be necessary to restrict accrual to patients who are suitable for, and have consented to, tumour and skin biopsies. Paired tumour biopsies are strongly recommended for all patients
* Patients must be ≥ 18 years of age.
* Patients must have an ECOG performance status of 0, 1, or 2.
* Presence of clinically and/or radiologically documented disease. All radiology studies must be performed within 28 days prior to registration (within 35 days if negative).

  * Phase I: patients do not need to have measurable disease
  * Phase I Expansion: patients must have measurable disease
* Previous Therapy

Cytotoxic Chemotherapy:

* Phase I: There is no limit to the number of prior regimens received.
* Phase I Expansion: Patients must have received at least one but no more than 3 regimens for advanced disease (Note: adjuvant anthracycline/taxane containing chemotherapy is considered an advanced regimen) Note: initially, there is no limitation to the use of prior platinumor PARPi containing regimens. During the expansion accrual may be limited to patients considered to be platinum naive, or platinum sensitive (no evidence of disease progression on or within 3 months of the last dose) or PARPi naïve or exposed. Sites will be informed at the time of the opening of the cohorts

Other Systemic Therapy:

• There is no limit to the number of prior therapies.

Patients must have recovered (to baseline or ≤ grade 1) from all reversible toxicity related to prior chemotherapy or systemic therapy and have adequate washout as follows:

Longest of one of the following:

* Two weeks,
* 5 half-lives for investigational agents,
* Standard cycle length of standard therapies.

Radiation:

Prior external beam radiation is permitted provided a minimum of 28 days (4 weeks) have elapsed between the last dose of radiation and date of registration. Exceptions may be made for low-dose, non-myelosuppressive radiotherapy after consultation with CCTG. Concurrent radiotherapy is not permitted.

Surgery:

Previous surgery is permitted provided that a minimum of 28 days (4 weeks) have elapsed between any major surgery and date of registration, and that wound healing has occurred.

* Lab Requirements Absolute neutrophils: ≥ 1.5 x 10^9/L Platelets: ≥ 100 x 10^9/L Bilirubin: ≤ 1.5 x ULN (upper limit of normal) AST/ALT: ≤ 2.5 x ULN ≤ 5.0 x ULN if patient has liver metastases Serum creatinine: ≤ 1.25 x ULN Creatinine clearance: ≥ 50 mL/min
* Women/men of childbearing potential must have agreed to use two effective contraceptive methods while on study and for 6 months after the last dose of CX5461.
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements.
* Patients must be accessible for treatment and follow up.
* Treatment is to begin within 2 working days of patient registration.

Exclusion Criteria:

- Other Malignancies

Phase I - Patients with other malignancies requiring concurrent anticancer therapy.

Phase I Expansion - Patients with a history of other malignancies, except:

* adequately treated non-melanomatous skin cancer,
* curatively treated in-situ cancer, or
* other solid tumours curatively treated at least 2 years prior to registration with no evidence of disease and not requiring concurrent anticancer treatment.

  * Patients with symptomatic brain metastases or spinal cord compression. Patients with asymptomatic brain/spinal cord metastasis who are not planned for radiation, or who have been treated and are stable off steroids (or on a decreasing dose) and anticonvulsants are eligible.
  * History of hypersensitivity to CX5461 or any excipient.
  * Patients with known photosensitivity disorders (xeroderma pigmentosa, porphyria etc). Patients who do not agree to use sunglasses and sun blocker (with SPF >30 to UVB and a high degree of protection against UVA) if exposed to sunlight during the course of the study and for 3 months after the last dose. Patients who plan to use sun beds or tanning booths during the course of the study and within 3 months after the last dose are not eligible.
  * Patients who have untreated and/or uncontrolled cardiovascular conditions documented within the last year:
* unstable angina,
* congestive heart failure,
* myocardial infarction,
* cardiac ventricular arrhythmias requiring medication,
* history of 2nd or 3rd degree atrioventricular conduction defects.

Patients who do not have untreated or uncontrolled cardiovascular conditions within the last year must have a LVEF ≥ 50%.

* Concurrent treatment with other investigational drugs or anti-cancer therapy.
* Patients with active or uncontrolled infections or with serious illnesses or medical conditions which would not permit the patient to be managed according to the protocol.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-06-13 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2023-01-18 (Actual)

PRIMARY OUTCOMES:
Confirm the recommended phase II dose and schedule of CX5461 in patients with solid tumours | 12 months

SECONDARY OUTCOMES:
Number and severity of adverse events in patients | 12 months
  To establish the safety and tolerability of CX5461 given intravenously to patients with solid tumours.
Assess pharmacokinetics of CX5461 | 12 months
  To determine the pharmacokinetics of CX5461 given intravenously to patients with solid tumours

CONTACTS AND LOCATIONS:
Overall Officials: Karen Gelmon, Study Chair — BCCA - Vancouver Cancer Centre; John Hilton, Study Chair — Ottawa Hospital Research Institute
Locations (3):
- Canada (3):
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hilton J, Gelmon K, Bedard PL, Tu D, Xu H, Tinker AV, Goodwin R, Laurie SA, Jonker D, Hansen AR, Veitch ZW, Renouf DJ, Hagerman L, Lui H, Chen B, Kellar D, Li I, Lee SE, Kono T, Cheng BYC, Yap D, Lai D, Beatty S, Soong J, Pritchard KI, Soria-Bretones I, Chen E, Feilotter H, Rushton M, Seymour L, Aparicio S, Cescon DW. Results of the phase I CCTG IND.231 trial of CX-5461 in patients with advanced solid tumors enriched for DNA-repair deficiencies. Nat Commun. 2022 Jun 24;13(1):3607. doi: 10.1038/s41467-022-31199-2. PMID 35750695
- [Derived] Xu H, Di Antonio M, McKinney S, Mathew V, Ho B, O'Neil NJ, Santos ND, Silvester J, Wei V, Garcia J, Kabeer F, Lai D, Soriano P, Banath J, Chiu DS, Yap D, Le DD, Ye FB, Zhang A, Thu K, Soong J, Lin SC, Tsai AH, Osako T, Algara T, Saunders DN, Wong J, Xian J, Bally MB, Brenton JD, Brown GW, Shah SP, Cescon D, Mak TW, Caldas C, Stirling PC, Hieter P, Balasubramanian S, Aparicio S. CX-5461 is a DNA G-quadruplex stabilizer with selective lethality in BRCA1/2 deficient tumours. Nat Commun. 2017 Feb 17;8:14432. doi: 10.1038/ncomms14432. PMID 28211448